CLINICAL TRIAL: NCT01131182
Title: An Open-Label, Randomized Naturalistic Study to Evaluate the Incidence of Hypoglycemia Comparing Sitagliptin With Sulfonylurea Treatment in Patients With Type 2 Diabetes During Ramadan Fasting
Brief Title: Study of Sitagliptin Treatment in Patients With Type 2 Diabetes During Ramadan (0431-263)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-263; 2010_538
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg administered orally daily as monotherapy or in combination with metformin over the Ramadan period.
  Interventions: Drug: Sitagliptin phosphate; Drug: Metformin
- Sulfonylurea (Active Comparator): Sulfonylurea administered orally daily as monotherapy or in combination with metformin over the Ramadan period.
  Interventions: Drug: Comparator: Sulfonylurea; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin phosphate — Sitagliptin 100 mg tablet administered orally once daily over the Ramadan period.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Comparator: Sulfonylurea — Sulfonylurea (glibenclamide, glimepiride, or gliclazide) administered orally daily over the Ramadan period as per physician's prescription
  Arms: Sulfonylurea
Drug: Metformin — Participants could continue pre-study metformin as concomitant therapy during the study.
  Other Names: Glucophage

SUMMARY:
This study will examine whether the incidence of hypoglycemia in patients fasting for Ramadan is lower when treated with sitagliptin as compared to sulfonylurea treatment.

DETAILED DESCRIPTION:
This study and NCT01340768 (MK-0431-262) have the same design but are conducted under separate protocols, in different countries, according to local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Muslim men and women with type 2 diabetes
* Participants who intend to fast during the month of Ramadan
* Participants who have been on a stable dose of sulfonylurea for at least three months

Exclusion Criteria:

* Participants with type 1 diabetes mellitus
* Pregnant or breast feeding women
* Participants with hypersensitivity or contraindication to dipeptidyl peptidase (DPP-4) treatment
* Participants on insulin
* Participants on any class of oral diabetic therapy other than sulfonylurea or metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2010-06-13 (Actual); Primary Completion 2010-11-04 (Actual); Study Completion 2010-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Al Sifri S, Basiounny A, Echtay A, Al Omari M, Harman-Boehm I, Kaddaha G, Al Tayeb K, Mahfouz AS, Al Elq A, Radican L, Ozesen C, Katzeff HL, Musser BJ, Suryawanshi S, Girman CJ, Davies MJ, Engel SS; 2010 Ramadan Study Group. The incidence of hypoglycaemia in Muslim patients with type 2 diabetes treated with sitagliptin or a sulphonylurea during Ramadan: a randomised trial. Int J Clin Pract. 2011 Nov;65(11):1132-40. doi: 10.1111/j.1742-1241.2011.02797.x. Epub 2011 Sep 27. PMID 21951832
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1147 participants enrolled in the study, 1066 participants were randomized to treatment.
Groups:
- Sitagliptin: Sitagliptin 100 mg administered orally daily over the Ramadan period
- Sulfonylurea: Sulfonylurea administered orally daily over the Ramadan period as per physician's prescription
Period: Overall Study
Arm/Group | Sitagliptin | Sulfonylurea
Started | 529 | 537
Completed | 513 | 521
Not Completed | 16 | 16
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 14 | 15
Not completed — Other Reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin: Sitagliptin 100 mg administered orally daily over the Ramadan period. All participants as treated population, n=507.
- Sulfonylurea: Sulfonylurea administered orally daily over the Ramadan period as per physician's prescription. All participants as treated population, n=514.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Sulfonylurea | Total
Number analyzed (Participants) | 507 | 514 | 1021
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11) | 55 (10) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 259 | 497
  Male | 269 | 255 | 524

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With at Least One Symptomatic Hypoglycemic Event
Description: Symptomatic hypoglycemic event was determined based on the participant's self-reported symptoms including faintness, headache, confusion, anxiety, sweating, tremor, palpitation, nausea, pallor, dizziness, hunger, and sudden behavioral change.
Time Frame: 30 days: first day of Ramadan (August 11) to last day of Ramadan (September 10)
Population: All participants as treated population consisted of all randomized participants who received at least one dose of study treatment and returned at least one completed diary card during the Ramadan period.
Measure: Number; unit: proportion of participants
Arm/Group | Sitagliptin | Sulfonylurea
Number analyzed (Participants) | 507 | 514
proportion of participants | 0.07 | 0.13
Statistical Analysis 1: Comparison: Sitagliptin vs Sulfonylurea; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — Assessed for relative risk using prior therapy (monotherapy or combination therapy) as a stratification factor

2. Secondary Outcome: Proportion of Participants With at Least One Symptomatic or Asymptomatic Hypoglycemic Event
Description: Hypoglycemic event was based on the participant's self-report and/or finger-stick blood glucose level. Symptomatic hypoglycemic symptoms included faintness, headache, confusion, anxiety, sweating, tremor, palpitation, nausea, pallor, dizziness, hunger, and sudden behavioral change.
Time Frame: 30 days: first day of Ramadan (August 11) to last day of Ramadan (September 10)
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Sitagliptin | Sulfonylurea
Number analyzed (Participants) | 507 | 514
Proportion of participants | 0.08 | 0.18

ADVERSE EVENTS:
Description: All participants as treated population consisted of all randomized participants who received at least one dose of study treatment and returned at least one completed diary card during the Ramadan period.
Arm/Group | Sitagliptin | Sulfonylurea
Serious Adverse Events (participants affected / at risk) | 0/507 | 3/514
Other Adverse Events (participants affected / at risk) | 34/507 | 68/514
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=507) | Sulfonylurea (N=514)
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=507) | Sulfonylurea (N=514)
Hunger (General disorders) | 13 | 35
Dizziness (Nervous system disorders) | 20 | 38
Headache (Nervous system disorders) | 25 | 44
Tremor (Nervous system disorders) | 7 | 34
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 19 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.